CLINICAL TRIAL: NCT02239367
Title: Electronic Depression Decision Aid for Nurses in Primary Care: Development and Implementation in a Diverse Low-Income Population
Brief Title: Depression Decision Aid: Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1401014663; P30MH085943 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Depression Decision Aid protocol (Experimental): The Depression Decision Aid protocol, integrated into the Electronic Health Record (EHR), is a streamlined adaptation of an in-person Shared Decision-Making intervention. Shared decision-making, in contrast to traditional medical decision-making, involves a collaborative process where patients discuss personal values and preferences and clinicians provide information to arrive at an agreed upon treatment decision. The focus of the intervention is to empower the elderly depressed primary care patients and help them efficiently arrive at a treatment decision that can be successfully implemented.
  Interventions: Behavioral: Depression Decision Aid

INTERVENTIONS:
Behavioral: Depression Decision Aid — The Depression Decision Aid protocol, integrated into the Electronic Health Record (EHR), is a streamlined adaptation of an in-person Shared Decision-Making intervention.
  Other Names: Shared Decision Making

SUMMARY:
The goal of this proposed pilot study is to test the feasibility and acceptability of a Depression Decision Aid (DDA) protocol integrated into the Electronic Health Record (EHR) and used by nurses with depressed ambulatory care patients. The Depression Decision Aid protocol is a streamlined adaptation of an in-person Shared Decision-Making (SDM) intervention, and its goal is to increase patient involvement in clinically appropriate treatment decision-making as a way of strengthening treatment engagement and outcomes. The protocol guides ambulatory care nurses in helping depressed patients (Patient Health Questionnaire-9 [PHQ-9] >10) develop informed treatment preferences through a process of education and values clarification. We will target patients in the general medical clinic, whether currently receiving depression treatment or not, because depression is highly prevalent but often poorly managed in this population.

DETAILED DESCRIPTION:
The aims of this project are to evaluate the acceptability and feasibility of an electronic Depression Decision Aid protocol with nurses and patients using questionnaire and administrative data.

One to two nurses will deliver the Decision Aid protocol to 40 low-income patients (aged 21 and over) scoring >10 via routine PHQ-9 screening. Consenting nurses will be assessed regarding their satisfaction with the protocol following its use with each patient subject. Nurse fidelity to the protocol will be evaluated via their documentation of protocol use in the EHR. Consenting patient subjects will be assessed at baseline; week 1 to determine their decision about depression treatment, satisfaction with the decision-making process; and week 12 to determine treatment initiation or change, treatment adherence, and depressive status. Medical records will also be examined for documentation of medication prescription and other depression treatments.

The study will test the following hypothesis concerning the Depression Decision Aid protocol:

1. Feasibility and Acceptability: a) At least 85% of each nurse's intervention sessions will meet fidelity standards via Electronic Health Record (EHR) data; b) Nurses will report high levels of satisfaction with the Decision Aid; c) Patients will report high levels of satisfaction with the decision-making process;

ELIGIBILITY:
Inclusion Criteria:

* 21 years and older
* Medical outpatient presenting to the Lincoln Hospital ambulatory care clinic or geriatric sub-specialty clinic
* Screen positive for depression (Patient Health Questionnaire-9 score of 10 or greater)

Exclusion Criteria:

* Presence of significant alcohol or substance abuse, psychotic disorder, or bipolar disorder
* High suicide risk
* Cognitive impairment: Mini Mental Status Exam (MMSE) score less than 24.
* Acute or severe medical illness (ie. delirium, metastatic cancer, decompensated cardiac, liver, or kidney failure, major surgery, stroke, or myocardial infarction during the three months prior to entry.
* Inability to speak English or Spanish
* Aphasia interfering with communication

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-13 (Actual)

PRIMARY OUTCOMES:
Use of Depression Decision Aid protocol | 12 weeks
  The number of nurse's intervention sessions based on Electronic Health Record data

SECONDARY OUTCOMES:
Satisfaction with the Decision Aid Measure | 12 weeks
  The Nurse Satisfaction Scale includes a measure of usefulness, clarity, ease of use, and feasibility in terms of timing when using the Decision Aid.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Raue, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Lincoln Hospital- the New York City Health and Hospitals Corporation (HHC), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No